CLINICAL TRIAL: NCT05317546
Title: Neurobehavioral Effects of Cannabidiol in Youth Alcohol Use Disorder
Brief Title: Cannabidiol in Youth Alcohol Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00119770
Record Dates: First submitted 2022-03-21; First posted 2022-04-08 (Actual); Results first posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cannabidiol, Then Placebo (Experimental)
  Interventions: Drug: Cannabidiol
- Placebo, Then Cannabidiol (Experimental)
  Interventions: Drug: Cannabidiol

INTERVENTIONS:
Drug: Cannabidiol — In counterbalanced order, 50 youth (ages 16-22) will receive 600mg of cannabidiol or placebo three hours before a neuroimaging and behavioral assessment paradigm, separated by an approximate 18-day washout period.
  Other Names: Placebo

SUMMARY:
The goal of this study is to test cannabidiol (CBD) as a potentially effective candidate medication for youth alcohol use disorder (AUD). To accomplish this goal, this study will use a randomized, double-blind, within-subjects crossover design. In counterbalanced order, 50 youth (ages 16-22) will receive 600 mg of CBD or placebo three hours before a neuroimaging and behavioral assessment paradigm. The total amount of time the participant will be in the study is approximately one month.

ELIGIBILITY:
Age 16 to 22. Does or does not drink alcohol.

Ages: 16 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kirkland AE, Browning BD, Meredith LR, Robertson E, Herring C, Tomko RL, Gray KM, Squeglia LM. The neural and psychophysiological effects of cannabidiol in youth with alcohol use disorder: A randomized controlled clinical trial. Neuropsychopharmacology. 2025 Sep;50(10):1482-1492. doi: 10.1038/s41386-025-02141-z. Epub 2025 Jun 11. PMID 40500407

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from September 2022 to April 2024, and data collection was completed in June 2024. Participants were recruited using a mix of approaches, including social media campaigns and in-person events. All participants completed a centralized intake process for youth substance use studies at the Medical University of South Carolina to determine eligibility before consenting for this specific study.
Pre-assignment Details: All participants that were eligible and enrolled in the study (N= 36) completed randomized to a group.
Groups:
- Cannabidiol, Then Placebo: In counterbalanced order, 19 youth (ages 17-22) were randomized to receive 600mg of cannabidiol before placebo three hours before a neuroimaging and behavioral assessment paradigm, separated by an approximate 18-day washout period.
- Placebo, Then Cannabidiol: In counterbalanced order, 17 youth (ages 17-22) were randomized to receive 600mg of placebo before cannabidiol three hours before a neuroimaging and behavioral assessment paradigm, separated by an approximate 18-day washout period.
Period: First Allocation
Arm/Group | Cannabidiol, Then Placebo | Placebo, Then Cannabidiol
Started | 19 | 17
Completed | 19 | 17
Not Completed | 0 | 0
Period: First Wash-Out Period
Arm/Group | Cannabidiol, Then Placebo | Placebo, Then Cannabidiol
Started | 19 | 17
Completed | 18 | 15
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2
Period: Second Allocation
Arm/Group | Cannabidiol, Then Placebo | Placebo, Then Cannabidiol
Started | 18 | 15
Completed | 18 | 15
Not Completed | 0 | 0
Period: Second Wash-out Period
Arm/Group | Cannabidiol, Then Placebo | Placebo, Then Cannabidiol
Started | 18 | 15
Completed | 18 | 14
Not Completed | 0 | 1
Period: Follow-Up
Arm/Group | Cannabidiol, Then Placebo | Placebo, Then Cannabidiol
Started | 18 | 14
Completed | 18 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were eligible and enrolled completed randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cannabidiol, Then Placebo | Placebo, Then Cannabidiol | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.4 (1.5) | 20.5 (1.8) | 20.5 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 16 | 34
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 17 | 14 | 31
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 17 | 36

OUTCOME MEASURES:

1. Primary Outcome: Concentrations of Glx (i.e., Glutamate + Glutamine)
Description: Using magnetic resonance spectroscopy and a within-subjects design, we measured Concentrations of Glx (i.e., glutamate + glutamine) levels in the anterior cingulate cortex in adolescents during cannabidiol (600mg) or placebo administration. Values provided are absolute values (mmol/kg) measured 3 hours after medication administration. Due to complexities of this method, "normal" levels of Glx are not known; thus, we cannot make conclusions about the meaning of "higher" or "lower" glutamate levels when comparing cannabidiol to placebo.
Time Frame: Changes 3 hours after administration of 600mg CBD vs. placebo
Measure: Mean (Standard Deviation); unit: mmol/kg
Groups:
- Cannabidiol (600mg): Outcomes when participants were given cannabidiol (600mg)
- Placebo: Outcomes when participants were given matched placebo
Arm/Group | Cannabidiol (600mg) | Placebo
Number analyzed (Participants) | 34 | 35
mmol/kg | 18.76 (0.98) | 18.57 (1.15)
Statistical Analysis 1: Comparison: Cannabidiol (600mg) vs Placebo; An a priori power analysis was conducted to ensure power to detect differences in neurometabolite levels in the dACC. Due to type of modeling, participants were included even if they did not complete the second medication allocation; Test type: Superiority — We used linear mixed effects models containing the main effect of medication (CBD vs. placebo), visit (visit 1 vs. visit 2), and sequence (CBD/placebo vs. placebo/CBD) with random intercepts. For 1H-MRS models, brain tissue composition [Gray Matter: Brain Matter or GM:BM defined as GM/(GM+WM)] was included as a covariate; p = 0.33, Mixed Models Analysis — alpha < 0.05; Adjusted for brain tissue composition

2. Primary Outcome: GABA+
Description: Using magnetic resonance spectroscopy and a within-subjects design, we measured GABA+ (GABA plus macromolecules) levels in the anterior cingulate cortex in adolescents during cannabidiol (600mg) or placebo administration. Values provided are absolute values (mmol/kg) measured 3 hours after medication administration. Due to complexities of this method, "normal" levels of GABA are not known; thus, we cannot make conclusions about the meaning of "higher" or "lower" GABA levels when comparing cannabidiol to placebo.
Time Frame: Changes 3 hours after administration of 600mg CBD vs. placebo
Measure: Mean (Standard Deviation); unit: mmol/kg
Arm/Group | Cannabidiol (600mg) | Placebo
Number analyzed (Participants) | 34 | 35
mmol/kg | 4.25 (0.26) | 4.22 (0.34)
Statistical Analysis 1: Comparison: Cannabidiol (600mg) vs Placebo; Due to type of modeling, participants were included even if they did not complete the second medication allocation; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.75, Mixed Models Analysis — alpha <0.05; Adjusted for brain tissue composition

3. Primary Outcome: Alcohol Cue Reactivity Neural Activation
Description: Assessing the change in neural reactivity to alcohol cues after each round of medication: Cannabidiol vs. placebo. Cue reactivity is a type of learned response which is observed in individuals who use substances (e.g., alcohol) and involves significant physiological reactions to presentations of substance-related stimuli (i.e., alcohol images) in comparison to neutral images (e.g., non-alcoholic beverages ) measured by BOLD (Blood Oxygen Level-Dependent response). ROIs were (left and right hemisphere): amygdala, caudate, insula, nucleus accumbens, and putamen. The mean Z-statistic within each ROI mask is reported. A Z-score of 0 represents the population mean (e.g., no activation), where higher absolute Z-scores indicate greater evidence of activation (positive or negative) in the ROI compared to baseline. Z-scores do not have inherent clinical thresholds. Higher Z-scores generally reflect stronger task-related BOLD signal changes.
Time Frame: Changes 3 hours after administration of 600mg CBD vs. placebo
Population: 33 participants had complete, usable data (n=3 dropped out before visit 2; n=1 without MRI data at visit 2; n= 1 with head motion at visit 1).
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Cannabidiol (600mg) | Placebo
Number analyzed (Participants) | 33 | 33
Z-score
  Anterior Cingulate Cortex | 1.02 (1.58) | 0.87 (1.37)
  Nucleus Accumbens (L) | 0.62 (0.85) | 0.35 (1.28)
  Nucleus Accumbens (R) | 0.53 (0.91) | 0.56 (1.26)
  Amygdala (L) | 0.66 (1.23) | 0.55 (0.92)
  Amygdala (R) | 0.68 (1.10) | 0.47 (1.09)
  Caudate (L) | 0.29 (1.00) | 0.24 (0.84)
  Caudate (R) | 0.51 (1.00) | 0.35 (1.11)
  Insula (L) | 0.10 (1.37) | 0.33 (1.24)
  Insula (R) | 0.12 (1.23) | 0.30 (1.24)
  Putamen (L) | 0.40 (1.16) | 0.42 (1.12)
  Putamen (R) | 0.42 (1.14) | 0.37 (1.16)
Statistical Analysis 1: Comparison: Cannabidiol (600mg) vs Placebo; Several studies have demonstrated that CBD can modulate resting-state or task-based BOLD signal under similar study design (acute dosing, 600 mg CBD) with sample sizes smaller than our sample. Due to the modeling, only participants with usable data from both medication allocation visits were included. Contrast of interest was alcohol beverages vs. non-alcohol beverages; Test type: Superiority; p > 0.05, Mixed Models Analysis

4. Primary Outcome: Heart Rate Variability
Description: All participants underwent an in vivo, olfactory alcohol cue exposure procedure. Participants smelled water followed by the participant's preferred beverage containing alcohol and apple juice in a counterbalanced order for three minutes each, with a three-minute rest period in between each liquid. The contents were poured into a cup in the participant's presence. During the task, electrocardiogram data were collected and used to create the heart rate variability (HRV) outcome related to the Sympathetic: Vagal ratio, which is the ratio of low-frequency to high-frequency power, derived from spectral HRV analysis. Higher values suggest increased sympathetic activity or reduced vagal activity.
Time Frame: Changes 2 hours after administration of 600mg CBD vs. placebo
Population: Some participants did not have usable data based on data quality markers.
Measure: Mean (Standard Deviation); unit: frequency ratio
Arm/Group | Cannabidiol (600mg) | Placebo
Number analyzed (Participants) | 32 | 32
frequency ratio | 0.84 (0.37) | 0.81 (0.41)
Statistical Analysis 1: Comparison: Cannabidiol (600mg) vs Placebo; We were not able to complete a power calculation for this task. We used linear mixed effects models, containing the main effect of medication (CBD vs. placebo), visit (visit 1 vs. visit 2), and sequence (CBD/placebo vs. placebo/CBD) and cue-by-medication interaction terms. Random intercepts were included to account for individual differences; Test type: Superiority; p = 0.82, Mixed Models Analysis

5. Primary Outcome: PhenX Toolkit Alcohol Urges Questionnaire
Description: All participants underwent an in vivo, olfactory alcohol cue exposure procedure. Participants smelled water followed by the participant's preferred beverage containing alcohol and apple juice in a counterbalanced order for three minutes each, with a three-minute rest period in between each liquid. The contents were poured into a cup in the participant's presence. After each beverage exposure, self-reported alcohol craving was collected via the PhenX Toolkit Alcohol Urges Questionnaire (AUQ). The AUQ consists of eight statements about the participant's feelings and thoughts about drinking as they are completing the questionnaire (i.e., right now). The participant was asked to respond to each statement about alcohol craving via a 7-item Likert scale ranging from "strongly disagree" to "strongly agree" with a scare range of 8 to 56 where higher scores represent higher alcohol craving.
Time Frame: Changes 2 hours after administration of 600mg CBD vs. placebo
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol (600mg) | Placebo
Number analyzed (Participants) | 34 | 35
score on a scale
  Alcohol Cue | 23.18 (11.73) | 21.40 (11.22)
  Apple Juice Cue | 18.56 (9.65) | 17.63 (10.26)
  Water Cue | 16.47 (7.64) | 15.50 (7.14)
  Baseline | 16.18 (7.30) | 14.94 (6.80)
Statistical Analysis 1: Comparison: Cannabidiol (600mg) vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.21, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: At least 36 days (18-days for the first wash-out period and 18-days for the second wash-out period before follow-up)
Description: Participants were asked about adverse events at every visit. Medication allocation visits (visit 1 and visit 2) adverse events were assessed by a medical clinician. At the follow-up visit (visit 3), they were assessed by study staff.
Groups:
- Cannabidiol (600mg): Adverse events assessed after the acute Cannabidiol (600mg) administration and washout period (~18 days).
- Placebo: Adverse events assessed after the acute placebo administration and washout period (~18 days).
Arm/Group | Cannabidiol (600mg) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/35
Other Adverse Events (participants affected / at risk) | 2/34 | 2/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cannabidiol (600mg) (N=34) | Placebo (N=35)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry Mouth (General disorders) | 1 (1) | 0 (0)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-11): https://cdn.clinicaltrials.gov/large-docs/46/NCT05317546/Prot_SAP_001.pdf
  • Informed Consent Form (2023-08-08): https://cdn.clinicaltrials.gov/large-docs/46/NCT05317546/ICF_000.pdf